CLINICAL TRIAL: NCT00455377
Title: Airway Inflammation in Cement Dust Exposed Workers
Brief Title: Lung Function and Airway Inflammation in Portland Cement Workers
Acronym: SPUTUM
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Rikshospitalet University Hospital (Other); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Anne Kristin M. Fell, MD, PhD, Sykehuset Telemark
Other Study IDs: STHF 5690.11, REK S-00166
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Airway Inflammation; Peripheral Blood Inflammation Markers; Cement Dust Exposure
Keywords: Cement dust exposure; Induced sputum; Airway inflammation; Peripheral blood inflammation markers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Induced sputum samples and blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to examine inflammation in the airways and in peripheral blood, in workers in a cement plant i Norway.

DETAILED DESCRIPTION:
OBJECTIVE: Former studies have presented conflicting data on the association between exposure to Portland cement dust and respiratory effects. Our goal is to examine inflammation in the airways and in peripheral blood in subjects exposed to cement-dust.

METHODS: All non smoking, dust exposed, workers from one department in the largest cement plant in Norway, are invited to participate. The workers will perform spirometry and induced sputum (IS) after a period of regular work with cement dust exposure, and again after a minimum of 5 days without exposure. Information on respiratory symptoms, allergy and former respiratory disease will be given on a self-reported questionnaire. IS was performed and processed as described by Pin et al. Differential cell counts will be carried out. Inflammatory markers in induced sputum and in peripheral blood will be measured. We want to use a crossover design were the cases are used as their own controls, but we will also include external controls.

ELIGIBILITY:
Inclusion Criteria:

* Cement dust exposure
* Non-smoker or ex-smoker >3 years

Exclusion Criteria:

* Infectious disease during the last 3 weeks
* Chronic airway disease

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers from Norways largest cement plant
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percentage of neutrophile cells in induced sputum | Before and after a period of exposure
  A significantly higher percentage of neutrophils was observed in induced sputum samples from cement production workers collected during an exposed period compared with a nonexposed period and compared with external controls.
Concentration of Interleukin 1beta in induced sputum | Before and after a period of exposure to cement production dust
  The concentration of Interleukin 1beta was higher in the sputum of workers during an exposed period than that of the office workers or the external controls.

CONTACTS AND LOCATIONS:
Overall Officials: Johny Kongerud, MD, Phd,, Study Chair — Department of respiratory medicine, Radiumhospitalet-Rikshospitalet Medical Centre, Oslo
Locations (1):
- Sykehuset Telemark, Skien, Telemark, Norway

REFERENCES:
- [Result] Fell AK, Sikkeland LI, Svendsen MV, Kongerud J. Airway inflammation in cement production workers. Occup Environ Med. 2010 Jun;67(6):395-400. doi: 10.1136/oem.2009.047852. Epub 2009 Oct 22. PMID 19854695